CLINICAL TRIAL: NCT04384471
Title: Patient Living With Type 1 Diabetes' Experience During the COVID-19 Pandemic in Quebec
Brief Title: Covid-19 Pandemic: Patients' Experience in T1D
Status: Completed | Type: Observational
Sponsor: McGill University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-1079
Record Dates: First submitted 2020-05-01; First posted 2020-05-12 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Type1diabetes; Covid19
Keywords: Patient reported outcomes; Type1diabetes; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People living with Type 1 Diabetes: People from all ages living with type 1 diabetes in the Province of Quebec
  Interventions: Other: Online survey

INTERVENTIONS:
Other: Online survey — Participants are invited to answer an online questionnaire including both close-ended and open-ended questions about their experience during this sanitary crisis

SUMMARY:
Given the current situation with COVID-19 declared pandemic on March 11, 2020 and the requirement for physical distancing and to limit social interactions, and for some, to quarantine, the investigators will survey patients living with type 1 diabetes (and their families, if they are <18 years) about their current experience with their diabetes management to understand their needs.

The primary objective is to describe the exposition and the impact of COVID-19 pandemic on type 1 diabetes. The investigators will recruit people with type 1 diabetes from all ages living in Quebec to answer a short online survey.

DETAILED DESCRIPTION:
Recruitment of people with type 1 diabetes will be done via an email sent to the participants in the BETTER registry who agreed to be contacted for other studies.

Participants of 18 years old and more will be invited to answer to the questionnaire (adult version of the questionnaires).

If the person with diabetes is aged < 18 years old, their parents will be invited to answer with them the survey ("parent" version of the questionnaire):

* Parents from the registry (PWT1D less than 14 y.o.) will receive the invitation email
* Participants of 14 to 18 years old who self-registered to the BETTER registry will receive an invitation email. They will be invited to complete the questionnaire with their parents. They will only have access to the "parent" version of questionnaire.

Advertising may be done through publicity on BETTER's social media (ie., Facebook, Instagram), via the BETTER monthly newsletter to increase awareness toward this research project. However the link to start the study will only be available in the email sent to the registry participants.

If people with type 1 diabetes not registered in BETTER want to participate in the present study, they will be instructed to self-register first to the registry and they will then receive a specific email to participate in the current study.

Data collection:

This will be a short online survey completed through an electronic software platform from Research Electronic Data Capture (REDCap) clinical software (English or French). The first question of the survey will be the consent form. Participants will be invited to answer the other questions only after having read the consent form and selecting 'Agree'. The consent form will also be available as a PDF document for download. The investigators have used this method in the past for the BETTER registry study. Participants will then confirm their eligibility.

The survey will include questions on acute complication (severe hypoglycemia and diabetic ketoacidosis); hypoglycemia frequency; hyperglycemia; ability to get diabetes supplies and to access diabetes care; impact of the pandemic situation on daily life activities (e.g., food insecurity, physical activity); impact on stress, anxiety and depression. The investigators will use the PHQ-9 scale for depression screening and the GAD7 scale for generalized anxiety among adult participants. The investigators will use the Short Mood and Feelings Questionnaire (SMFQ) for child and adolescent. The version used is the own that has been adapted to be completed by parents . The SMFQ was developed for use in epidemiological studies of depression in children and adolescents.

If participants show a certain level of distress, as reflected by the PHQ9 questionnaire score (≥ 10) or the SMFQ score (≥ 8), they will receive an automated email with resources that they can contact.

For PWT1D, socio-demographic information (e.g., age, ethnicity and education) and diabetes history (e.g., diabetes duration, complications) will be retrieved from the BETTER registry. Data from the registry and from this specific questionnaire will be linked using 3 identification information: the email address, the date of birth and the sex. The investigators have used this methodology for the SUPPORT study.

Analysis: The investigators will use demographic information already available on the BETTER registry. This will be a descriptive analysis. Continuous data will be reported as means with standard deviations (median and interquartile range if data are skewed). Categorical data will be reported as proportions. The investigators will do regression analysis to explore the effect of the COVID-19 pandemic duration on the patients' experience.

Thematic analysis will be performed for the free text. Content will be coded and concepts will be categorized into different themes by two researchers.

Sample size:

Based on an estimated number of 70 000 PWT1D in Quebec, a sample size of 384 completed questionnaire was calculated with an error margin of 5%, a confidence interval of 95% and a distribution of answers of 50%, A 50% distribution was used because it is impossible to predict answers; this proportion corresponds to the scenario with the larger sample size needed. Sample size was calculated using Raosoft.

Importance of this study: This study will inform about the major issues experienced by patients living with diabetes. The anxiety and added stress may lead to dysregulated blood sugars and deteriorations in their physical and mental well-being. Accesses to health care services are limited. This study will inform on the support needed by patients with type 1 diabetes during this pandemic to avoid or limit negative consequences. This may help to advocate for more remotely accessible resources for patients.

ELIGIBILITY:
Inclusion criteria:

* Having type 1 diabetes
* Living in Quebec
* Having took part in the BETTER registry (www.type1better.com)

Exclusion criteria:

-Not understanding French or English

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: -People living with type 1 diabetes in Quebec and are registered to the BETTER registry.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Self-reported acute diabetes complication | Since March 11, 2020
  Severe hypoglycemia and diabetic ketoacidosis

SECONDARY OUTCOMES:
Self-reported hypoglycemia | Last 7 days
  In the last week, how many episodes of hypoglycemia did you have? Answer based on the following definition of hypoglycemia: measured blood sugar levels lower than 4.0 mmol/L and/or common symptoms [shaking, sweating, anxiety, confusion, difficulty concentrating, nausea, or other symptoms] and/or disappearance of symptoms with carbohydrate intake.
Ability to get diabetes supplies and to access diabetes care | Since March 11, 2020
  Since the start of the COVID-19 pandemic (March 11), have you had difficulty getting a hold of any of the following diabetes supplies Scale: 1- no difficulties at all to 7- I could not get any supplies i) Blood glucose meter ii) Blood glucose meter strips iii) Insulin iv) Glucagon v) Ketone strips vi) Continuous glucose monitor sensors or related supplies vii) Insulin pump supplies viii) Alcohol wipes
Concern about not having access to diabetes supplies and to access diabetes care | Since March 11, 2020
  Since the start of the COVID-19 pandemic (March 11), are you worried about access to any of the following diabetes supplies? Scale: 1- not at all worried to 7- I am very worried i) Blood glucose meter ii) Blood glucose meter strips iii) Insulin iv) Glucagon v) Ketone strips vi) Continuous glucose monitor sensors or related supplies vii) Insulin pump supplies viii) Alcohol wipes
Impact of the pandemic situation on daily life activities | Since March 11, 2020
  Two questions on food security
  One question on physical activity
Impact on stress, anxiety and depression for adults participants | Last 2 weeks
  PHQ-9 scale for depression screening and the GAD7 scale for generalized anxiety among adult participants.
Impact on stress, anxiety and depression for children and adolescents | Last 2 weeks
  Short Mood and Feelings Questionnaire (SMFQ) for children and adolescent.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie Brazeau, PhD, Principal Investigator — McGill University
Locations (1):
- Institut de Recherches Cliniques de Montréal, Montreal, Quebec, Canada